CLINICAL TRIAL: NCT03308435
Title: Effect of Transfemoral Transcatheter Aortic Valve Replacement (TF-TAVR) on Emotional Status, Quality of Life, Frailty and Inflammation and Their Interactions
Brief Title: Effect of TF-TAVR on Emotional Status, Quality of Life, Frailty and Inflammation
Status: Terminated | Type: Observational
Why Stopped: futility
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dirk von Lewinski, Assoc. Prof., Medical University of Graz
Other Study IDs: 29-371 ex 16/17
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Stenosis; Clinical Trial; Depression; Frail Elderly Syndrome; Inflammation
MeSH Terms: conditions — Aortic Valve Stenosis; Depression; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and blood cells will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Geriatric assessment — the assessment includes functional tests (hand grip strength, SPPB (Short Physical Performance Battery)) and questionaires Euro-QoL 5D, LUTS, GDS, ADL, iADL, dietary recall).
Diagnostic Test: Psychiatric assessment — Psychiatric assessments includes HAMD-17 as well as Beck depression inventory, hospital anxiety and depression scale, SF36, PTSS-10
Diagnostic Test: Inflammatory assessment — analysis will include arginase, ADMA, SDMA, homoarginine, aminoacids + metabolites, tryptophan, kynurenine, kynurenine acid, cortisol, ACTH, Metanephrine, myeloperoxidase,
Diagnostic Test: Cardiological assessment — ECG, echocardiography

SUMMARY:
Aortic valve stenosis (AS) shows high and increasing prevalence in Western civilizations and leads to high morbidity and mortality. 15 years ago Alain Cribier performed the first catheter-based transfemoral aortic valve replacement at the University of Rouon. This historical step initiated a dramatic shift in the treatment of AS with more than 50% of patients being treated interventionally instead of the surgical approach, today.

Comorbidities are major determinants of cardiovascular events and clinical outcome in aortic valve stenosis but little is known about psychiatric comorbidities or frailty in these patients. Data from our group suggest an inflammatory trigger for depression and potentially other psychiatric diseases and aortic valve stenosis as well as aortic valve replacement are associated with considerable changes in the inflammatory state of the patients. However, no study has prospectively examined the interaction of these inflammatory markers and mood disorders, yet. In addition, frailty is a key aspect of many of TAVR patients clinically, however, scientifically there is only emerging data with half of all PubMed-indexed publications being less than 18 months old and clinical use of various scores still under discussion.

The " Effect of interventional aortic valve replacement on emotional status, quality of life, frailty and inflammation"-study is designed to fill these gaps in evidence. It will be a prospective epidemiological cohort study to recruit 102 patients with symptomatic severe aortic valve stenosis within 18 months. All of these patients will undergo standardized cardiologic, psychiatric and frailty assessment as well as a sophisticated laboratory analysis focussing on the inflammatory state. The study aims to integrate these interdisciplinary findings to optimize patient treatment.

DETAILED DESCRIPTION:
Aortic valve stenosis (AS) shows a high prevalence in Western civilizations with an increasing incidence and is associated with high morbidity and mortality. AS is a degenerative disease and therefore the main reason for the increasing prevalence is the higher proportion of elderly patients in western societies. Untreated symptomatic AS is characterized by severe morbidity with mainly dyspnea, orthopnea and reduced exercise capacity. In addition, AS has a very high mortality (50-90% in 2 years), most often due to lung edema as a result of increased afterload of the left ventricle. So far, there is no medical treatment available improving mortality in these patients. For decades, the only known therapy has been surgical aortic valve replacement (SAVR), having shown a dramatic reduction in mortality. However, many of the patients suffering from AS are octogenarians or even older and also suffer from multiple comorbidities. Thus, many of these patients are considered inoperable using a surgical approach. Exactly 15 years ago Alain Cribier performed the first catheter-based transfemoral aortic valve replacement at the University of Rouon. This historical step initiated a dramatic shift in the treatment of AS with more than 50% of patients being treated interventionally instead of the surgical approach, today.

Comorbidities are major determinants of cardiovascular events and clinical outcome in aortic valve stenosis but little is known about psychiatric comorbidities or frailty in these patients. Data from our group suggest an inflammatory trigger for depression and potentially other psychiatric diseases and aortic valve stenosis as well as aortic valve replacement are associated with considerable changes in the inflammatory state of the patients. However, no study has prospectively examined the interaction of these inflammatory markers and mood disorders, yet. In addition, frailty is a key aspect of many of TAVR patients clinically, however, scientifically there is only emerging data with half of all PubMed-indexed publications being less than 12 months old and clinical use of various scores still under discussion.

The " Effect of interventional aortic valve replacement on emotional status, quality of life, frailty and inflammation"-study is designed to fill these gaps in evidence. It will be a prospective epidemiological cohort study to recruit 102 patients with symptomatic severe aortic valve stenosis within 18 months. All of these patients will undergo standardized cardiologic, psychiatric and frailty assessment as well as a sophisticated laboratory analysis focussing on the inflammatory state. The study aims to integrate these interdisciplinary findings to optimize patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic aortic valve stenosis
* Planned elective transcatheter aortic valve replacement
* Willingness and ability to provide signed informed consent (IC) form prior to participation in any study-related procedures

Exclusion Criteria:

* Disease reducing life expectancy to < 1 year
* Severe immune-system modulating or -affecting disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve stenosis scheduled for transfemoral aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Aortic valve area | 6 months
  valve area as measured calculated by doppler echocardiography

SECONDARY OUTCOMES:
HAMD-17 (Hamilton) | 6 months
  questionaire score
BDI-II | 6 months
  Beck depression inventory score
SF-36 | 6 months
  short form-36 questionaire
PTSS-10 | 6 months
  Post traumatic syndrome scale-10
Euro-QoL5D | 6 Months
  Quality of life questionaire
hand grip strenght test | 6 months
  hand grip strenght test
BIA | 6 Months
  Bioelectrical impedance analysis
kynurenine acid | 6 months
  inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Schmidt, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided
data will be shared with cooperating colleagues of the geriatric, psychiatric and laboratory departments